CLINICAL TRIAL: NCT03308708
Title: Prophylactic Norepinephrine Infusion for Spinal-induced Hypotension
Brief Title: Norepinephrine for Spinal-induced Hypotension
Acronym: NE in spianl
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NE_spinal
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Spinal Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- NE group (Experimental)
  Interventions: Drug: Norepinephrine infusion

INTERVENTIONS:
Drug: Norepinephrine infusion — Norepinephrine infusion (5miclml) is immediately started after spinal anesthesia. Rate starts at 30 ml/h and modified according to hemodynamic state
  Arms: NE group

SUMMARY:
Norepinephrine (NE) infusion is used prophylactically to counteract the vasodilator effect of spinal anesthesia. prophylactic use of NE infusion is expected to decrease bouts of hypotension, vomiting and increase patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective surgery under spinal anesthesia

Exclusion Criteria:

* ischemic heart disease uncontrolled hypertension

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
incidence of hypotension | intraoperative
  intraoperative decrease of patient blood pressure by more than 20% from its basal reading

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Manşūrah, Dkahleya, Egypt